CLINICAL TRIAL: NCT02296151
Title: Evaluation of Treatment Factors in the Management of Chronic Iliotibial Band Syndrome in Female Distance Runners.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Janine SieuNarine-McKay, Dr. Janine McKay, University of British Columbia
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: H13-01816
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Iliotibial Band Syndrome
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Placebo Comparator): Four iliotibial band stretches; to be completed 3 days per week.
  Interventions: Other: iliotibial band stretches
- Group B (Active Comparator): Four conventional hip exercises (Hip abductor, gluteus medius strengthening); to be completed 3 days per week.
  Interventions: Other: Gluteus medius strengthening
- Group C (Experimental): Four conventional hip exercises progressed during the 8-weeks, totalling 16 exercises over the 8-week period (Hip abductor, gluteus medius strengthening). Exercises to be completed 3 days per week.
  Interventions: Other: Gluteus medius strengthening

INTERVENTIONS:
Other: Gluteus medius strengthening — Hip abductor, gluteus medius strengthening
  Arms: Group B; Group C
Other: iliotibial band stretches — Iliotibial band stretches
  Arms: Group A

SUMMARY:
The primary objective of this study is to determine if a more specific exercise routine that incorporates a progressive hip stability program will help to rehabilitate the hip and reduce symptoms of iliotibial band syndrome more than conventional hip exercises. Three different exercises interventions will be compared to determine its effectiveness in reducing pain, improving function and returning subjects to running symptom free. Secondary objective for this study is to establish an intervention program for female runners with this injury. There will be three treatment arms and participants will be randomly assigned to one of three groups: Group A- control (stretching), group B (conventional hip exercises and group C (experimental treatment- specific progressive hip exercises).

DETAILED DESCRIPTION:
The gluteus medius muscle is part of a muscle group called the hip abductor muscles. The gluteus medius originates at the dorsal ilium (uppermost, largest bone of the pelvis) below the iliac crest and inserts at the top outside surfaces of the greater trochanter (top of the thigh bone). It is the major abductor of the thigh (moves the leg away from the midline of the body). The anterior fibres rotate the hip internally and the posterior fibres rotate the hip externally. Based on the anatomy and function of this muscle, the gluteus medius plays a major role in the mechanics of running. Research has shown that runners with iliotibial band syndrome have been shown to have weakness in this muscle. Most conventional exercises that have been research have been exercises that focus on only activation of this muscle in an unloaded position (non-weightbearing). Group B of this study will focus on those exercises that have been researched. Group C will be the experimental group in which we will begin with the conventional exercises and progress the exercises from a floor (unloaded) position to a more dynamic functional position (standing). This will be geared towards running specific exercises. We would like to know if there will be a difference in how fast symptoms reduce and strength gains occur and at what rate.

ELIGIBILITY:
Inclusion Criteria:

1. Female between the ages of 19-45 years;
2. Have been diagnosed or been affected by ITBS (pain on the outside of the knee) for no less than 3 months;
3. A distance runner averaging a minimum of 15 Km per week of road running;

Exclusion Criteria:

1. Have previous history of knee surgery or knee trauma to the affected side;
2. Have been diagnosed with any other knee pathology such as patellofemoral pain syndrome, degenerative joint disease, chondromalacia patella, tendinitis or tendinopathy in the affected knee;

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Hip dynamometer strength | 8-weeks
  Hip dynamometer strengthening will be measured biweekly for the 8-week period

SECONDARY OUTCOMES:
Y-balance test | Measured pre and post 8-week study
  The Y-balance test kit is designed to measure quality of movement and function in three different movement planes.
Single leg mini squat | Measured pre and post 8-week study
  The single leg mini squat will be used to assess quality of movement.

OTHER OUTCOMES:
Numeric pain scale | Measured weekly for the duration of the 8-week study
  This is subjective rating scale 0-10. Participants will rate their pain weekly.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rick Celebrini, PhD, PT, Study Chair — Chief sport officer- Fortius sport & health; Dr. Michael Hunt, MSc MPT PhD, Study Chair — Assistant Professor (UBC)- Department of Physical Therapy
Locations (1):
- Optimal Performance Clinic, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Agre JC, Magness JL, Hull SZ, Wright KC, Baxter TL, Patterson R, Stradel L. Strength testing with a portable dynamometer: reliability for upper and lower extremities. Arch Phys Med Rehabil. 1987 Jul;68(7):454-8. PMID 3606371
- [Result] Beers A, Ryan M, Kasubuchi Z, Fraser S, Taunton JE. Effects of Multi-modal Physiotherapy, Including Hip Abductor Strengthening, in Patients with Iliotibial Band Friction Syndrome. Physiother Can. 2008 Spring;60(2):180-8. doi: 10.3138/physio.60.2.180. Epub 2008 Oct 10. PMID 20145781
- [Result] Birnbaum K, Siebert CH, Pandorf T, Schopphoff E, Prescher A, Niethard FU. Anatomical and biomechanical investigations of the iliotibial tract. Surg Radiol Anat. 2004 Dec;26(6):433-46. doi: 10.1007/s00276-004-0265-8. PMID 15378277
- [Result] Devan MR, Pescatello LS, Faghri P, Anderson J. A Prospective Study of Overuse Knee Injuries Among Female Athletes With Muscle Imbalances and Structural Abnormalities. J Athl Train. 2004 Sep;39(3):263-267. PMID 15496997
- [Result] Fairclough J, Hayashi K, Toumi H, Lyons K, Bydder G, Phillips N, Best TM, Benjamin M. The functional anatomy of the iliotibial band during flexion and extension of the knee: implications for understanding iliotibial band syndrome. J Anat. 2006 Mar;208(3):309-16. doi: 10.1111/j.1469-7580.2006.00531.x. PMID 16533314
- [Result] Fredericson M, Cookingham CL, Chaudhari AM, Dowdell BC, Oestreicher N, Sahrmann SA. Hip abductor weakness in distance runners with iliotibial band syndrome. Clin J Sport Med. 2000 Jul;10(3):169-75. doi: 10.1097/00042752-200007000-00004. PMID 10959926